CLINICAL TRIAL: NCT00552604
Title: Randomised, Double-blind, Placebo-controlled Phase III Trial to Determine the Efficacy and Safety of a Standardised Oral Extract of Cannabis Sativa for the Symptomatic Relief of Muscle Stiffness and Pain in Multiple Sclerosis.
Brief Title: MUltiple Sclerosis and Extract of Cannabis (MUSEC) Study
Acronym: MUSEC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to recruitment problems / based on recommendation of Independent Review Board
Sponsor: Institut fur Klinische Forschung, Germany (Other)
Collaborators: Weleda AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-01; EUDRA-CT No.; 2005-005263-29
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Muscle Spasticity
Keywords: multiple sclerosis; muscle stiffness; spasticity; pain; treatment; cannabinoids
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cannabis extract (delta-9-THC 2.5mg, CBD 1.25 mg per capsule), flexible dosing between 5 mg and 25 mg THC/d, administered twice daily
  Interventions: Drug: standardized cannabis extract
- 2 (Placebo Comparator): matching placebo capsules, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: standardized cannabis extract — Cannabis extract (delta-9-THC 2.5mg, CBD 1.25 mg per capsule), flexible dosing between 5 mg and 25 mg THC/d, administered twice daily
  Arms: 1
Drug: Placebo — Matching placebo capsules, twice daily
  Arms: 2

SUMMARY:
Study Objectives: To determine the efficacy and safety of a standardised extract of Cannabis sativa given orally 2 times daily as compared to placebo for the relief of muscle stiffness and pain in multiple sclerosis for a period of 12 weeks.

Study Patients: 400 patients with multiple sclerosis (age 18-64, stable disease during previous 6 months, ambulatory or not, antispasticity medication and physiotherapy stabilised ≥ 30 days) with experiencing muscle stiffness ≥ 4 on a 11-point numerical Likert scale at baseline.

Study treatment:

Group 1: Cannabis extract (delta-9-THC 2.5mg, CBD 1.25 mg per capsule), flexible dosing between 5 mg and 25 mg THC/d, administered twice daily, additionally to previous antispasticity and analgesic medication.

Group 2: Matched placebo, twice daily, additionally to previous antispasticity and analgesic medication.

Treatment Schedule: Start dose 5 mg THC/d, individual dose titration with increase of 5 mg THC every 3 days, maximal total daily dose 25 mg THC, administered as 2 equal doses based on tolerability. Treatment duration: 12 weeks.

Study sites: 20 neurological clinics in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Diagnosis of MS according to McDonald criteria.
* Current muscle stiffness ≥ 4 on a 11-point categorical rating scale.
* On-going troublesome muscle stiffness for at least 3 months.
* Stable disease for the previous 6 months.
* Antispasticity medication and physiotherapy stabilised for the last 30 days.
* Patients may be ambulatory or not.
* Age 18-64.

Exclusion Criteria:

* Immunosuppressants which may affect spasticity (including corticosteroids and interferon but ex-cluding azathioprine) taken currently or in previous 30 days
* Past or present history of psychotic illness.
* Open/infected pressure sores or other source of chronic infection.
* Significant fixed tendon contractures.
* Severe cognitive impairment such that the patient is unable to provide informed consent.
* History of clinically important renal, cardiovascular or neurol. diseases (apart from MS).
* Malignancy within the past 2 years.
* Cannabinoids taken currently or in previous 30 days.
* Positive qualitative urinary test on cannabinoids at screening visit. (In this case a patient will be allowed to repeat the test at a second screening visit later.)
* Known hypersensitivity to cannabinoids.
* Current drug abuse, including alcohol abuse.
* Laboratory parameters outside the following limits:

Creatinine > 3x upper limit of normal Bilirubine > 3x upper limit of normal Transaminases > 5 x upper limit of normal

* Anticipated immunisations within the 12 weeks of trial participation.
* Other problems likely to make participation difficult at the discretion of the neurologist.
* Women who are pregnant, lactating or not using adequate contraception.
* Participation in other treatment studies currently or within the previous month.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness: 11-point numerical Likert scale | 12 weeks

SECONDARY OUTCOMES:
Change in pain: 11-point numerical Likert scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John J Zajicek, Prof., Principal Investigator — Peninsula Medical School, University of Plymouth, UK
Locations (1):
- Peninsula Medical School, Plymouth, Plymouth, United Kingdom

REFERENCES:
- [Derived] Zajicek JP, Hobart JC, Slade A, Barnes D, Mattison PG; MUSEC Research Group. Multiple sclerosis and extract of cannabis: results of the MUSEC trial. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1125-32. doi: 10.1136/jnnp-2012-302468. Epub 2012 Jul 12. PMID 22791906